CLINICAL TRIAL: NCT06096142
Title: Prospective, Randomized, Controlled, Multicenter Study of the Solaris DE Endoprosthesis in the Treatment of Venous Outflow Stenosis or Occlusion in Hemodialysis Patients
Brief Title: The Solaris DE Endoprosthesis for the Treatment of AV Access Stenosis or Occlusion
Acronym: DEScover
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Scitech Produtos Medicos Ltda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SCI-SD-001
Record Dates: First submitted 2023-10-17; First posted 2023-10-23 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Venous Stenosis; Venous Occlusion; Chronic Renal Failure
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- AVF Treatment (Experimental): Participants on dialysis via AV fistula will be treated with percutaneous transluminal angioplasty (PTA) followed by Solaris DE implantation.
  Interventions: Device: Solaris DE
- AVF Control (Sham Comparator): Participants on dialysis via AV fistula will be treated with percutaneous transluminal angioplasty (PTA) alone.
  Interventions: Device: PTA
- AVG Treatment (Experimental): Participants on dialysis via AV graft will be treated with percutaneous transluminal angioplasty (PTA) followed by Solaris DE implantation.
  Interventions: Device: Solaris DE

INTERVENTIONS:
Device: Solaris DE — Percutaneous Transluminal Angioplasty (PTA) followed by Solaris DE implantation in the treated vessel.
  Arms: AVF Treatment; AVG Treatment
Device: PTA — Percutaneous Transluminal Angioplasty (PTA) in the treated vessel alone.
  Arms: AVF Control

SUMMARY:
The goal of this clinical trial is to demonstrate the safety and efficacy of Solaris DE Endoprosthesis in the treatment of stenosis or occlusion within the outflow circuit of the dialysis access including arteriovenous (AV) fistula and synthetic AV graft.

Participants will be treated with Solaris DE Endoprosthesis. Researchers will compare the treatment with investigational product to Percutaneous Transluminal Angioplasty (PTA) alone within the AV fistula cohort in order to demonstrate superiority of Solaris DE.

DETAILED DESCRIPTION:
This is a prospective, randomized (1:1), controlled, multicenter study to investigate the safety and efficacy of the Solaris DE Endoprosthesis in the treatment of hemodialysis patients with stenosis or occlusion of the venous outflow circuit. The study population includes two cohorts:

* AVF cohort: participants presenting an arteriovenous fistula (AVF) stenosis or occlusion of the peripheral venous outflow circuit, including the cephalic arch, will be randomized 1:1 between treatment with the test device (Solaris DE) or standard treatment by Percutaneous Transluminal Angioplasty (PTA) alone);
* AVG cohort: participants with an arteriovenous graft (AVG) presenting stenosis or occlusion at the graft vein anastomosis or juxta-anastomosis or at the segment of the prosthesis exit circuit, will be treated with the test device (Solaris DE) only.

ELIGIBILITY:
Inclusion Criteria:

* The participant has a mature AV Fistula (AVF) or Graft (AVG) in the arm created ≥ 30 days before the initial procedure and is in use for dialysis therapy
* The participant has clinical and/or hemodynamic evidence of a venous outflow obstruction or AV fistula or graft dysfunction. The stenotic lesion is ≥ 50%, with a maximum length of 8 cm and a vessel diameter from 4.0 mm to 9.0 mm
* The participan provides written informed consent prior to any study-specific procedure
* The participan is willing to undergo all follow-up evaluations according to the specified schedule over 24 months

Angiographic Inclusion Criteria:

* The target lesion originates ≥ 3 cm from the cannulation segment (needling zone)
* The target lesion is located:

  1. In one arm (including the cephalic arch) in a participant with AVF, and not in the cannulation segment, OR
  2. In the anastomosis or juxta-anastomosis in a participant with AVF (a juxta-anastomosis is defined as a location where the stent crosses the venous anastomosis)
* The target lesion includes a de novo stenotic lesion or restenosis
* The target lesion is ≥ 5 cm from the arterial anastomosis
* The target lesion has ≥ 50% stenosis according to the operator's visual judgment
* The reference vessel diameter of the target lesion is between 4.0 mm and 9.0 mm by the operator's visual judgment
* Single or multiple target lesions measuring ≤ 8 cm in total length by the operator's visual judgment
* Single or multiple target lesions should be covered by a single stent or multiple overlapping stents, provided they are treated as a single lesion with a maximum length of 8 cm
* Successful target lesion pre-dilatation is defined as crossover of the guidewir resulting in full expansion of the pre-dilatation balloon
* The participant has up to 1 (one) non-target lesion in the venous outflow circuit requiring intervention in the initial procedure. The non-target lesion must be at least 10 cm away from the target lesion. The non-target lesion can only be treated with standard PTA alone
* Does not have stent implanted or it has been in the access circuit for ≥ 30 days since placement and patent with ≤ 30% stenosis and located ≥ 5 cm from the target lesion
* The non-target lesion must be successfully treated at the time of the initial procedure (success measured as ≤30% residual stenosis and no complications).

Exclusion Criteria:

* Pregnant, breastfeeding or with intention to become pregnant in the next year
* The participant has any major endovascular or surgical procedure planned (including in the access circuit) within 30 days of the initial procedure
* It was not possible to pre-dilate the lesion to be treated with Solaris DE
* Planned surgical revision of the access site
* Known or suspected infection of the hemodialysis access site, systemic infection and/or sepsis
* Patients on immunosuppressive therapy
* Known active coagulopathy or bleeding diathesis
* Known hypersensitivity to nickel titanium alloy, contrast or sirolimus
* Contraindication to antiplatelet, anticoagulant or thrombolytic therapies
* Known allergy to contrast agents or medications administered to perform endovascular intervention that cannot be adequately premedicated
* Life expectancy of less than 12 months
* Has a stent or endoprosthesis located anywhere in the AV access circuit that is not patent (> 30% stenosis) or implanted < 30 days
* The participant's hemodialysis access is expected to be abandoned within 6 months
* The participantis is enrolled in another trial involving an investigational product (pharmaceutical, biological or medical device)

Angiographic Exclusion Criteria:

* The target lesion is located inside an endoprosthesis
* Target lesion treatment would involve the cannulation segment (needling zone)
* The target lesion is < 5 cm from the arterial anastomosis
* Evidence of an aneurysm, pseudoaneurysm or acute thrombus (i.e. one that has been treated ≤ 15 days) within the target lesion
* The target lesion is, and/or Solaris DE would be placed anywhere:

  1. Through the elbow
  2. In the cannulation segment (needling zone)
  3. Inside any part of a pre-existing stent or endoprosthesis (apart from an access arteriovenous graft)
  4. Lower extremity
  5. Non-synthetic graft
* The target lesion is located in such a way that the insertion of a stent would result in a "kink" area that requires a stent bridge between the Solaris DE and an existing stent or stent graft
* The individual has more than 1 (one) non-target lesion (≥ 50% stenosis) that requires intervention in the initial procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-08-30 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
Safety Events | 30 days
  Percentage of participants without any safety events affecting the access or venous outflow circuit and resulting in new intervention, hospitalization or death (not including stenosis or thrombosis).
Target Lesion Primary Patency (TLPP) | 6 months
  Percentage of participants without restenosis or clinically indicated target lesion revascularization or thrombosis.

SECONDARY OUTCOMES:
Target Lesion Primary Patency (TLPP) | 12 and 24 months
  Percentage of participants without restenosis or clinically indicated target lesion revascularization or thrombosis.
Assisted Target Lesion Primary Patency (aTLPP) | 1, 6, 12 and 24 months
  Percentage of participants without uncorrectable occlusion of the target lesion since the procedure.
Access Circuit Primary Patency (ACPP) | 1, 6, 12 and 24 months
  Percentage of participants without any new venous outflow circuit intervention, thrombosis or access abandonment since the procedure.
Cumulative Patency (CP) | 1, 6, 12 and 24 months
  Percentage of participants without the access circuit abandonment since the procedure.
Procedure and device-related complications | 1, 6, 12 and 24 months
  Complication rates related to the procedure and device involving the access circuit.

CONTACTS AND LOCATIONS:
Overall Officials: Leonardo O Harduin, MD, Principal Investigator — Hospital Universitário Pedro Ernesto - Universidade do Estado do Rio de Janeiro (HUPE-UERJ); Fábio H Rossi, MD, Principal Investigator — Instituto Dante Pazzanese de Cardiologia; Leonardo C Almeida, MD, Principal Investigator — Hospital Ana Nery; Thiago A Almeida, MD, Principal Investigator — Afya Hospital Dia LTDA; Douglas E T Cavalcanti, MD, Principal Investigator — Real Hospital Português de Beneficência em Pernambuco; Guilherme C Santos, MD, Principal Investigator — Hospital das Clínicas da UFMG/EBSERH
Locations (6):
- Brazil (6):
  - Hospital Ana Nery, Salvador, Estado de Bahia
  - Afya Hospital Dia LTDA, Brasília, Federal District
  - Hospital das Clínicas da UFMG/EBSERH, Belo Horizonte, Minas Gerais
  - Real Hospital Português de Beneficência em Pernambuco, Recife, Pernambuco
  - Hospital Universitário Pedro Ernesto - UERJ, Rio de Janeiro, Rio de Janeiro
  - Instituto Dante Pazzanese de Cardiologia, São Paulo, São Paulo

IPD SHARING:
Plan to Share IPD: No